CLINICAL TRIAL: NCT03788876
Title: Neuromuscular Electrical Stimulation After Lung Transplantation: Randomized Clinical Trial.
Brief Title: Neuromuscular Electrical Stimulation After Lung Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180497
Record Dates: First submitted 2018-11-27; First posted 2018-12-28 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lung Transplantation; Electric Stimulation; Clinical Trial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular electrical stimulation (Active Comparator): The NMES training will be applied once a day (30 minutes of application per session with an increase of one minute every two days and reduction in the OFF time), until the discharge from the ICU. The patient will continue with the application also in the Hospitalization Units of HCPA and Irmandade da Santa Casa de Misericórdia de Porto Alegre until discharge and the protocol of physiotherapy by the physiotherapists of HCPA twice a day that will consist in exercises for bronchial hygiene, exercises for pulmonary reexpansion and exercises of passive mobilization.
  Interventions: Other: Neuromuscular electrical stimulation; Other: Conventional care
- Conventional care (Sham Comparator): The protocol of physiotherapy by the physiotherapists of HCPA and Irmandade da Santa Casa de Misericórdia de Porto Alegre twice a day that will consist in exercises for bronchial hygiene, exercises for pulmonary reexpansion and exercises of passive mobilization.
  Interventions: Other: Conventional care

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — The NMES training will be applied once a day (30 minutes of application per session with an increase of one minute every two days and reduction in the OFF time), until the discharge from the ICU. The patient will continue with the application also in the Hospitalization Units of HCPA and Irmandade da Santa Casa de Misericórdia de Porto Alegre until discharge.
  Arms: Neuromuscular electrical stimulation
Other: Conventional care — Physiotherapy protocol will be performed by HCPA and Irmandade da Santa Casa de Misericórdia de Porto Alegre physiotherapists twice a day, which will consist of exercises for bronchial hygiene, exercises for pulmonary reexpansion, and passive mobilization exercises.

SUMMARY:
Pulmonary transplantation aims to increase patient survival and quality of life in relation to functional aspects. It is observed that the decrease in muscle mass and pulmonary changes are some complications that can be found in the post-transplant patient due to immobility. Thus, Neuromuscular Electrical Stimulation (NMES) rehabilitation is of paramount importance for the recovery of the individual, both in the functional aspects, and in the minimization in the time of hospitalization.The objective of this study was to evaluate the effects of NMES on the thickness and strength of the quadriceps femoris muscle, pulmonary function, endothelial function, functional capacity, muscle biochemical markers, arterial blood gas analysis and water balance of patients after lung transplantation through a randomized clinical trial. Patients will be randomized into two groups: EENM group: will receive the application of NMES associated with physiotherapy and control group: who will receive only the physiotherapy protocol of the Hospital of Clinics of Porto Alegre (HCPA) and Irmandade da Santa Casa de Misericórdia de Porto Alegre.

DETAILED DESCRIPTION:
Pulmonary transplantation aims to increase patient survival and quality of life in relation to functional aspects. It is observed that the decrease in muscle mass and pulmonary changes are some complications that can be found in the post-transplant patient due to immobility. Thus, NMES rehabilitation is of paramount importance for the recovery of the individual, both in the functional aspects, and in the minimization in the time of hospitalization.The objective of this study was to evaluate the effects of NMES on the thickness and strength of the quadriceps femoris muscle, pulmonary function, endothelial function, functional capacity, muscle biochemical markers, arterial blood gas analysis and water balance of patients after lung transplantation through a randomized clinical trial. Patients will be randomized into two groups: EENM group: will receive the application of NMES associated with physiotherapy and control group: who will receive only the physiotherapy protocol of the HCPA. The NMES training will be applied once a day (30 minutes of application per session, increasing one minute every two days and reducing the OFF time), until the discharge of the Intensive Care Unit (ICU). The patient will continue with the application also in the Hospitalization Units of the HCPA and Irmandade da Santa Casa de Misericórdia de Porto Alegre until the hospital discharge. The following outcomes will be evaluated: thickness and strength of the quadriceps muscle, pulmonary function, endothelial function, functional capacity, mobility, muscle biochemical markers, arterial blood gas analysis, water balance and length of stay in the ICU, time and success of weaning from invasive mechanical ventilation and survival rate through medical records analysis.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral and Unilateral lung transplant;
* After extubation of invasive mechanical ventilation up to 48 hours for stable patients;
* After extubation of invasive mechanical ventilation up to 72 hours for those who are present in the instability;
* Chronic obstructive pulmonary disease
* Cystic fibrosis
* Fibrotic pulmonary idiopathic

Exclusion Criteria:

* Skin lesions at the electrode placement points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Femoral quadriceps muscle thickness | three weeks
  Performed through a Portable Ultrasound System (VIVID i®, GE) with a linear arrangement probe (60 mm, 7.5 MHz - VIVID i®, GE).
Muscle quadriceps muscle quality Evaluation of muscle quality through ultrasound images | three weeks
  Performed through a Portable Ultrasound System (VIVID i®, GE) with a linear arrangement probe (60 mm, 7.5 MHz - VIVID i®, GE).

SECONDARY OUTCOMES:
Muscle Strength - Scale Medical Research Council (MRC) | three weeks
  The MRC score is obtained by evaluating 12 muscle groups in the upper extremities (wrist extensors, elbow flexors, and shoulder abductors) and lower limbs (dorsal ankle flexors, knee extensors, and hip flexors). Each muscle group will be given a score between 0 (complete paralysis) and 5 (normal strength), and the total score can range from 0 to 60 points.
Dynamometry | three weeks
  Dynamometry = handgrip test
Sit and stand up | three weeks
  At the starting signal the subject will have to get up until standing and returning to a sitting position. The subject will be encouraged to perform 10 consecutive repetitions in the shortest possible time interval.
30 meter walk test | three weeks
  Evaluates walking speed for six minutes
Spirometry | three weeks
  Evaluates lung function
Blood Markers | three weeks
  Evaluates markers of muscle injury.
Hydric balance | three weeks
  Through patient records
length of stay in the ICU | three weeks
  Through patient records
Length of stay in invasive mechanical ventilation | three weeks
  Through patient records
Time of weaning from invasive mechanical ventilation | three weeks
  Through patient records
Survival Rate | three weeks
  Through patient records
Success of weaning from invasive mechanical ventilation | three weeks
  Through patient records

CONTACTS AND LOCATIONS:
Overall Officials: Graciele Sbruzzi, Principal Investigator — Hospital of Clinics of Porto Alegre
Locations (2):
- Brazil (2):
  - HCPA, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No